CLINICAL TRIAL: NCT00842127
Title: Genetic Polymorphism of Drug Transporters in OROS-Methylphenidate Treatment in Children and Adolescents With Attention Deficit Hyperactivity Disorder(ADHD)
Brief Title: Genetic Polymorphism and OROS-Methylphenidate Treatment in Attention Deficit Hyperactivity Disorder(ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Ki-Hwan Yook, Bundang CHA hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEPOROM; A030001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Methylphenidate; ADHD; Multidrug resistance(MDR)polymorphism; OROS methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: OROS-methylphenidate (Concerta) — dose: 18mg, 27mg, 36mg, 45mg, 54mg/day, po duration: 8 weeks
  Other Names: Concerta

SUMMARY:
The purpose of this study is to examine whether genetic polymorphisms in drug transporters were associated with the side effects of OROS-methylphenidate medication in attention deficit/hyperactivity disorder(ADHD).

DETAILED DESCRIPTION:
20 to 30% of children with attention deficit/hyperactivity disorder(ADHD) do not respond or could not tolerate methylphenidate treatment. Drug transporters such as multidrug resistant proteins(MDR) plays important role in the clearance of psychotropic drugs and their metabolites from brain tissue. It suggested that methylphenidate was a P-glycoprotein(encoded by MDR1 gene)substrate and showed inhibitory effects on the P-glycoprotein efflux function. Single nucleotide polymorphisms(SNP)in the MDR1 gene were analyzed in children and adolescents with OROS-methylphenidate treatment. The hypothesis is that MDR1(ABCB1) polymorphisms are associated with the side effects of OROS-methylphenidate.

ELIGIBILITY:
Inclusion Criteria:

* ADHD
* Must be able to swallow a capsule

Exclusion Criteria:

* Pervasive developmental disorder
* Mental retardation
* Psychotic disorder
* Bipolar disorder
* Suicidality
* Neurological disorder
* Concurrent psychiatric treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Barkley side effects rating scale | weeks 1, 2,4,8

SECONDARY OUTCOMES:
ADHD rating scale-Korean version; Clinical Global Impressions (CGI) of Severity and Improvement (CGI-S and CGI-I) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Hwan Yook, MD,PhD, Principal Investigator — Department of psychiatry CHA university college of medicine
Locations (1):
- Bundang CHA hospital, Seongnam, Kyonggi-do, South Korea